CLINICAL TRIAL: NCT01106378
Title: Cynergy - The CYPHER-NEVO Registry. An Observational Registry, to Evaluate the Safety and Performance of the NEVO™ Sirolimus-eluting Coronary Stent in Routine Clinical Practice, and to Compare Its Safety and Performance With the CYPHER Select® Plus Sirolimus-eluting Coronary Stent (SES)
Brief Title: Cynergy: the CYPHER-NEVO Registry
Acronym: CYNERGY
Status: Terminated | Type: Observational
Why Stopped: Early termination of patient enrollment based on business decision
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Hans-Peter Stoll, MD, PhD, Cordis Corporation
Other Study IDs: EC09-02
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; drug-eluting stents; sirolimus-eluting coronary stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NEVO™ Sirolimus-eluting Coronary Stent System.: Subjects treated during routine clinical practice with the NEVO™ Sirolimus-eluting Coronary Stent System and diagnosed with acute STEMI for primary intervention and/or diabetes mellitus and/or multi vessel disease.
- CYPHER Select® Plus Coronary Stent: Subjects treated during routine clinical practice with the CYPHER Select® Plus Coronary Stent System and diagnosed with acute STEMI for primary intervention and/or diabetes mellitus and/or multi vessel disease

SUMMARY:
The purpose of this registry is to compare the safety and the performance of the NEVO™ Sirolimus-eluting Coronary Stent, once commercially available, to the CYPHER Select® Plus Sirolimus-eluting Coronary Stent in complex subjects presenting with acute STEMI for primary intervention, diabetes mellitus or multi vessel disease. The second purpose of this registry is to evaluate the safety and performance of the NEVO™ Sirolimus-eluting Coronary Stent, once commercially available and the CYPHER Select® Plus Sirolimus-eluting Coronary Stent in complex subjects diagnosed with acute STEMI for primary intervention, diabetes mellitus and/or multi vessel disease.

The data will be collected from subjects treated with commercially available product and following routine clinical practice. Uniform, complete and accurate data will be collected on the subject's medical history, peri-procedurally, during the index hospitalization, and during follow-up.

DETAILED DESCRIPTION:
The CYPHER Select® Plus Sirolimus-eluting Coronary Stent (SES) is a balloon-expandable intracoronary 316L stainless steel stent with a coating that consists of a blend of Sirolimus and polymers.

Sirolimus is a potent immunosuppressive agent which has been proven to prolong graft survival in many animal models of transplantation. Sirolimus prevents both proliferation and migration of smooth muscle cells (in vivo and in vitro) in graft and balloon injury models. Furthermore, Sirolimus has been shown to be effective in reducing restenosis and the need for repeat revascularization while demonstrating superior efficacy measures such as angiographic late loss and binary restenosis.

The NEVO™ Sirolimus-eluting Coronary Stent is a cobalt-chromium alloy stent platform that incorporates two unique features: reservoir technology, and a bioresorbable polymer which prevents initial contact between the polymer and the vessel wall and chronic polymer exposure. This design minimized initial tissue exposure to polymer, and also enables polymer resorption within approximately three months.

ELIGIBILITY:
Inclusion criteria:

- Subjects treated in routine clinical practice with a NEVO™ Sirolimus-eluting Coronary Stent once commercially available, or a CYPHER Select® Plus Sirolimus-eluting Coronary Stent and diagnosed with acute STEMI for primary intervention and/or diabetes mellitus and/or multi vessel disease.

Exclusion criteria:

* In case, during the index procedure, the subject was treated with a stent other than the CYPHER Select® Plus Sirolimus-eluting Coronary Stent or the NEVO™ Sirolimus-eluting Coronary Stent or a mix of the CYPHER Select® Plus SES and NEVO™ SES
* In case, during the index procedure, the subject was treated with other therapy (e.g. balloon angioplasty, cutting balloons, directional coronary atherectomy, excimer laser, rotational atherectomy, thrombectomy, etc.) in segments not ultimately treated with a CYPHER Select® Plus SES or NEVO™ SES.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects treated in routine clinical practice with a NEVO™ Sirolimus-eluting Coronary Stent,once commercially available, OR a CYPHER Select® Plus Sirolimus-eluting Coronary Stent and diagnosed with acute STEMI for primary intervention and/or diabetes mellitus and/or multi vessel disease.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority comparison of Target Lesion Failure (TLF) in the NEVO group to the CYPHER group in subjects with acute STEMI, diabetes mellitus or multi vessel disease. | 12 months follow-up post-procedure
  TLF: composite clinical endpoint of cardiac death (death that cannot be attributed to a non-cardiac cause), target vessel-related MI and clinically-driven target lesion revascularization in the NEVO group compared to the CYPHER group.

SECONDARY OUTCOMES:
TLF in the NEVO and the CYPHER group | Discharge, 1, 6, and 24 months follow-up post-procedure
  TLF: composite clinical endpoint of cardiac death (death that cannot be attributed to a non-cardiac cause), target vessel-related MI and clinically driven target lesion revascularization
Prescription and compliance patterns and impact of dual antiplatelet therapy (DAPT) duration on the incidence of the composite endpoint of all death, all MI and all revascularization, its individual components,stent thrombosis (ST) and major bleeding. | Duration throughout the study
Clinically driven Target Lesion Revascularization (TLR) defined as repeat PCI or CABG to the target lesion | Hospital discharge, 1, 6, 12 and 24 months follow-up post-procedure
Clinically driven Target Vessel Revascularization (TVR) defined as repeat PCI or CABG to the target vessel | Hospital discharge, 1, 6, 12 and 24 months follow-up post-procedure
Composite endpoint of all death, all MI, all revascularization and its individual components | Hospital discharge, 1, 6, 12 and 24 months follow-up post-procedure
Incidence of ARC (Academic Research Consortium) defined (definite, probably, possible and the composite of definite and probable) early and late and very late stent thrombosis | Hospital discharge, 1,6, 12 and 24 months follow-up post-procedure
Major bleeding complications | Hospital discharge, 1, 6, 12 and 24 months follow-up post-procedure.
Stroke that persists >24 hours | Hospital discharge, 1, 6, 12 and 24 months follow-up post-procedure.
  Stroke (cerebrovascular accident or CVA) defined as sudden onset of vertigo, numbness, dysphasia, weakness, visual field defects, dysarthria or other focal neurological deficits due to vascular lesions of the brain such as hemorrhage, embolism, thrombosis, or rupturing aneurysm, that persists >24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Philip Urban, MD, Principal Investigator — Clinique La Tour; Expedito Ribeiro, MD, Principal Investigator — Instituto do Coracão do Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo; Seung Jung Park, MD, Principal Investigator — Asan Medical Center
Locations (3):
- Instituto do Coracão do Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil
- Asan Medical Center, Seoul, South Korea
- Clinique La Tour, Meyrin, Switzerland